CLINICAL TRIAL: NCT06992024
Title: Electroacupuncture Combined With Paclitaxel Protein-bound and PD-1 Antibody for Second-line Treatment of HER2 Negative, pMMR/MSS Advanced Gastric Cancer: a Prospective, Open-labeled, Single-arm, Phase Ⅱ Clinical Trial
Brief Title: Electroacupuncture Combined With Paclitaxel Protein-bound and PD-1 Antibody for Second-line Treatment of HER2 Negative, pMMR/MSS Advanced Gastric Cancer
Acronym: EAPPA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250554
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Electroacupuncture Combined With Paclitaxel Protein-bound and PD-1 Antibody for Second-line Treatment of HER2 Negative, pMMR/MSS Advanced Gastric Cancer
Keywords: electroacupuncture; paclitaxel protein-bound; PD-1 antibody; HER2 negative, pMMR/MSS advanced gastric cancer
MeSH Terms: interventions — Taxes

STUDY DESIGN:
Intervention Model Description: Electroacupuncture Combined With Paclitaxel Protein-bound and PD-1 Antibody for Second-line Treatment of HER2 Negative, pMMR/MSS Advanced Gastric Cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EA+Chemo+IO (Experimental): Electroacupuncture (EA) Combined With Paclitaxel Protein-bound (Chemo) and PD-1 Antibody (IO) for Second-line Treatment of HER2 Negative, pMMR/MSS Advanced Gastric Cancer. Electroacupuncture stimulates specific acupoints（dense-sparse wave，30min）d0, d1, d7, d8 + Paclitaxel Protein-bound (125mg/m2) d1, d8 + PD-1 Antibody (not limited to specific drugs，dosages should be calculated according to corresponding drug instructions) d1, Q3W.
  Interventions: Combination Product: Electroacupuncture Combined With Paclitaxel Protein-bound and PD-1 Antibody

INTERVENTIONS:
Combination Product: Electroacupuncture Combined With Paclitaxel Protein-bound and PD-1 Antibody — Electroacupuncture (EA) Combined With Paclitaxel Protein-bound (Chemo) and PD-1 Antibody (IO) for Second-line Treatment of HER2 Negative, pMMR/MSS Advanced Gastric Cancer. Electroacupuncture stimulates specific acupoints（dense-sparse wave，30min）d0, d1, d7, d8 + Paclitaxel Protein-bound (125mg/m2) d1, d8 + PD-1 Antibody (not limited to specific drugs，dosages should be calculated according to corresponding drug instructions) d1, Q3W. If the diseases are well controlled after 6 cycles, maintenance treatment, namely Electroacupuncture stimulates specific acupoints（dense-sparse wave，30min）d0, d1 + PD-1 Antibody (not limited to specific drugs，dosages should be calculated according to corresponding drug instructions) d1, Q3W, will be continually conducted until the diseases progress.

SUMMARY:
There are several basic findings in the previous studies: The levels of renin and aldosterone in the blood of cancer patients vary greatly among individuals, and the baseline levels of some patients are relatively higher than others; The elevated levels of renin and aldosterone in the blood are positively correlated with the higher malignancy, drug resistance and progression of gastric cancer; Electroacupuncture stimulation of relevant acupoints can effectively down-regulate the levels of renin and aldosterone in the blood; Electroacupuncture stimulation of relevant acupoints can effectively activate the function of the immune system.

Based on these findings, the present clinical trial aim to evaluated the efficacy and safety of electroacupuncture combined with chemotherapy and PD-1 Antibody for the treatment of specific type of gastric cancer.

DETAILED DESCRIPTION:
The number of new cases of gastric cancer ranks fifth among all cancers worldwide, and the number of deaths from gastric cancer ranks fourth. In 2020, the number of global deaths from gastric cancer was close to 770,000. Gastric cancer is a common malignant tumor in China. In 2020, the number of new cases ranked second and the number of deaths ranked third. The number of new cases was approximately 480,000, accounting for 43.9% of the global total, and the number of deaths was about 370,000, accounting for 48.6% of the global total. Moreover, gastric cancer with clinical stages III-IV accounted for about 60%. For HER2-negative advanced gastric cancer, chemotherapy based on platinum-based, fluorouracil and paclitaxel has been regarded as the standard treatment approach in the past few decades. However, the effect of chemotherapy is extremely limited, and the objective response rate of first-line treatment is only 40%-50%. With the clinical application of immune checkpoint inhibitors, the treatment strategies for gastric cancer have undergone revolutionary changes. However, the objective response rate of immune checkpoint inhibitor monotherapy for advanced gastric cancer is only 11%-15% [1]. This means that most patients find it difficult to benefit from monotherapy with immune checkpoint inhibitors. Chemotherapy combined with immune checkpoint inhibitors is a feasible method to overcome drug resistance. A phase III, multicenter international study KEYNOTE 859 demonstrated that the combination of immune checkpoint inhibitor pembrolizumab (a PD-1 monoclonal antibody) and chemotherapy as first-line treatment for locally advanced unresectable or metastatic HER2-negative gastric cancer could significantly prolong the median overall survival time (OS) of patients compared with placebo combined with chemotherapy (P < 0.0001). Maintain a better quality of life score, and Chinese patients can benefit from pembrolizumab combined with chemotherapy (median OS 15.9 months, objective response rate (ORR) 69%) [2]. Therefore, in December 2023, pembrolizumab was approved in China for the first-line treatment of patients with locally advanced unresectable or metastatic HER2-negative gastric or gastroesophageal junction adenocarcinoma in combination with fluorouracil and platinum-based chemotherapy. Her2-negative, complete mismatch repair gene/microsatellite stable (pMMR/MSS) advanced gastric cancer is a difficulty in the treatment of gastric cancer. Especially, there are no large-scale phase III clinical research data for second-line treatment after the progression of first-line treatment. According to the latest version of the Chinese CSCO diagnosis and treatment guidelines, for this type of patients, chemotherapy ± immune checkpoint inhibitors (such as PD-1 monoclonal antibodies, etc.) are recommended as the first-line treatment. After the progression of the first-line treatment, the second-line treatment is recommended as either monotherapy with paclitaxel or monotherapy with irinotecan or paclitaxel combined with the anti-vascular targeted drug ramoxifumab. Considering the economic situation of patients in the real world, Most patients can only receive monotherapy, and the control effect of monotherapy on the disease is extremely limited. There is no large-scale clinical research data on whether chemotherapy combined with PD-1 monoclonal antibody can bring benefits to patients in the second-line treatment of advanced gastric cancer.

Electroacupuncture therapy, as an important treatment method in traditional Chinese medicine, has been widely proven to improve various diseases by regulating the levels of multiple hormones in the body and regulating the immune function. In previous studies, our research group and other research groups found that electroacupuncture stimulation of specific acupoints can significantly down-regulate the levels of blood renin and aldosterone, and the effect is particularly obvious for patients whose baseline levels of blood renin and aldosterone are higher than the normal range [3, 4]. The levels of renin and aldosterone in the blood have been confirmed to be positively correlated with the malignancy degree and progression rate of gastric cancer [5].

Based on the above previous findings, this study proposes a new treatment strategy for HER2-negative advanced gastric cancer patients with pMMR/MSS who progressed after first-line chemotherapy with fluorouracil and platinum-based regimens ±PD-1 monoclonal antibody treatment, and adopts the second-line electroacupuncture + Paclitaxel Protein-bound +PD-1 monoclonal antibody regimen. The efficacy and safety of this regimen are intended to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following study enrollment criteria:

Age ≥18 years old and ≤75 years old; Pathology and imaging confirmed advanced gastric cancer with HER2 negative and pMMR/MSS; Progression after first-line chemotherapy with fluorouracil and platinum-based regimens and ±PD-1 monoclonal antibody treatment, second-line treatment is planned; The ECOG score is 0-2; Life expectancy > 3 months; Willing and able to accept follow-up until death or the end of the study or the termination of the study; The hematological function is normal (platelets > 80×10^9/L; White blood cells > 3×10^9/L; Neutrophils > 1.5×10^9/L; Serum bilirubin ≤1.5 times the upper limit of normal value (ULN), transaminase ≤5 times ULN; There was no ascites, the coagulation function was normal, and the albumin was ≥30g/L; The Child-Push classification of liver function is grade A; Serum creatinine is less than the upper limit of the normal value (ULN), or the calculated creatinine clearance rate is > 50ml/min (using the Cockcroft-Gault formula) ;

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the study:

The primary tumor recurred; Severe arterial embolism or ascites; There is a tendency to bleed or coagulation disorder; Hypertensive crisis or hypertensive encephalopathy; Severe and uncontrollable systemic complications such as infections or diabetes; Clinical severe cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (within 6 months before enrollment), hypertension that remains uncontrolled after appropriate drug treatment, unstable angina pectoris, congestive heart failure (NYHA grades 2-4), and arrhythmias requiring drug treatment; Have suffered from or whose physical examination shows central nervous system diseases (such as primary brain tumors, epilepsy that cannot be controlled by standard treatment, any history of brain metastases or strokes); Have suffered from other malignant tumors in the past five years (excluding basal cell carcinoma of the skin and/or carcinoma in situ of the cervix after radical resection); Be allergic to any drug in the study; Pregnant and lactating women; There are any other diseases, functional disorders caused by metastatic lesions, or suspected disorders found during physical examinations, suggesting that there may be contraindications to the use of the studied drug or putting the patient at high risk of treatment-related complications; Unable or unwilling to comply with the research protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The proportion of patients whose tumors have shrunk to the expected value and can persist until the expected minimum time limit requirement according to the RECIST criteria

SECONDARY OUTCOMES:
Disease control rate (DCR) | 2 years
  The proportion of patients whose tumors were classified as CR (complete response), PR (partial response), and SD (stable disease) according to the RECIST criteria
Progression-free survival time (PFS) | 2 years
  The time from the start of randomization to tumor progression or death
PFS rate | 2 years
  The proportion of patients who did not experience tumor progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Han Z, Cheng S, Dai D, Kou Y, Zhang X, Li F, Yin X, Ji J, Zhang Z, Wang X, Zhu N, Zhang Q, Tan Y, Guo X, Shen L, Peng Z. The gut microbiome affects response of treatments in HER2-negative advanced gastric cancer. Clin Transl Med. 2023 Jul;13(7):e1312. doi: 10.1002/ctm2.1312. PMID 37381590
- [Background] Rha SY, Oh DY, Yanez P, Bai Y, Ryu MH, Lee J, Rivera F, Alves GV, Garrido M, Shiu KK, Fernandez MG, Li J, Lowery MA, Cil T, Cruz FM, Qin S, Luo S, Pan H, Wainberg ZA, Yin L, Bordia S, Bhagia P, Wyrwicz LS; KEYNOTE-859 investigators. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for HER2-negative advanced gastric cancer (KEYNOTE-859): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Nov;24(11):1181-1195. doi: 10.1016/S1470-2045(23)00515-6. Epub 2023 Oct 21. PMID 37875143
- [Background] Lee HS, Kim JY. Effects of acupuncture on blood pressure and plasma renin activity in two-kidney one clip Goldblatt hypertensive rats. Am J Chin Med. 1994;22(3-4):215-9. doi: 10.1142/S0192415X94000279. PMID 7872233
- [Background] Zhang M, Zhu Y, Wang J, Li Y, Hua Z. Association between acupuncture and grade 1 hypertension: A systematic review and meta-analysis. Complement Ther Clin Pract. 2022 Nov;49:101649. doi: 10.1016/j.ctcp.2022.101649. Epub 2022 Aug 7. PMID 35963138
- [Background] Sugimoto M, Yamaoka Y, Shirai N, Furuta T. Role of renin-angiotensin system in gastric oncogenesis. J Gastroenterol Hepatol. 2012 Mar;27(3):442-51. doi: 10.1111/j.1440-1746.2011.06964.x. PMID 22114933